CLINICAL TRIAL: NCT03910231
Title: The Role of Vasopressin Antagonism on Renal Sodium Handling
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jonathan S. Williams, MD, MMSc, Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2012P000638
Record Dates: First submitted 2019-04-09; First posted 2019-04-10 (Actual); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: vasopressin receptor; renal sodium excretion
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Intervention Model Description: Randomized, placebo-controlled, double-blinded, parallel arm clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Blinding to investigator, participant and study staff. Randomization assignment and blinding provided by Investigational Drug Services
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Tolvaptan Oral Tablet
- 15mg Tolvaptan (Experimental): 15mg Tolvaptan
  Interventions: Drug: Tolvaptan Oral Tablet
- 30mg Tolvaptan (Experimental): 30mg Tolvaptan
  Interventions: Drug: Tolvaptan Oral Tablet

INTERVENTIONS:
Drug: Tolvaptan Oral Tablet — Tolvaptan, to block V2R

SUMMARY:
Vasopressin has primarily been considered to be a water and osmosis regulating hormone that mediates its effects on renal aquaporin channels. Recent data suggest that vasopressin, through its V2 receptor, may also modulate sodium homeostasis. The purpose of this human physiology study was to test whether antagonism of the V2R alters urine sodium excretion in normal healthy volunteers.

DETAILED DESCRIPTION:
Vasopressin's potential roles in maintaining normal volume homeostasis are expanding. While previous data support the concept that vasopressin's primary role is in mediating water homeostasis, recent data suggest that vasopressin, through its V2 receptor, may also modulate sodium homeostasis. This effect occurs via activation of the epithelial sodium channel (ENaC). These studies document that vasopressin via activation of the V2 receptor, not only reduces free water excretion but also sodium excretion. These data suggest that blocking this receptor under the right circumstances and in the right population may be effective in modulating hypertension in humans: specifically a V2 receptor antagonist may be effective in treating some individuals that have salt-sensitive hypertension. The current proposal will test in normal human subjects the proof of principle of the above stated hypothesis, and to assess the best markers to determine such an effect. It is important to perform studies with strict environmental control in a clinical research center because of the variability of environmental factors that can create confusion in interpreting data (dietary sodium, activity, body posture, diurnal variation, ambient temperature, sleep-wake cycle, etc.).

The overall program objective is to determine if a vasopressin V2 antagonist will be an effective treatment for salt-sensitive hypertension and if so, what subtype. The object of this specific proposal is to determine the effect of a selective V2 antagonist on sodium handling in normal subjects.

ELIGIBILITY:
Inclusion Criteria:

* - Blood pressure <130/85 mmHg and >100/50 mmHg
* Normal laboratory values for (see "Normal Values" table):
* Complete blood count
* Serum creatinine, sodium, potassium, glucose, liver enzymes
* Urinalysis
* ECG

Exclusion Criteria:

* - Alcohol intake >12 oz per week
* Tobacco or recreational drug use
* History of coronary disease, diabetes, hypertension, stroke, kidney disease, or illness requiring overnight hospitalization in the past 6 months
* Any prescription medication or herbal medication use except oral contraceptive or multivitamin
* Pregnancy or current breastfeeding
* First degree relative with hypertension, diabetes, stroke, renal or cardiac disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2015-02-01 (Actual)

PRIMARY OUTCOMES:
Acute intravenous saline response | 6 hours
  Urine sodium excretion measured in response to saline infusion

SECONDARY OUTCOMES:
Dietary salt response | 6 days
  Cumulative sodium excretion measured in response to dietary salt loading

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Williams, MD, MMSc, Principal Investigator — Brigham and Women's Hospital

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: October 2019 for 1 year

REFERENCES:
- [Background] Stockand JD. Vasopressin regulation of renal sodium excretion. Kidney Int. 2010 Nov;78(9):849-56. doi: 10.1038/ki.2010.276. Epub 2010 Aug 25. PMID 20736986
- [Background] Bankir L, Bichet DG, Bouby N. Vasopressin V2 receptors, ENaC, and sodium reabsorption: a risk factor for hypertension? Am J Physiol Renal Physiol. 2010 Nov;299(5):F917-28. doi: 10.1152/ajprenal.00413.2010. Epub 2010 Sep 8. PMID 20826569
- [Background] Blanchard A, Frank M, Wuerzner G, Peyrard S, Bankir L, Jeunemaitre X, Azizi M. Antinatriuretic effect of vasopressin in humans is amiloride sensitive, thus ENaC dependent. Clin J Am Soc Nephrol. 2011 Apr;6(4):753-9. doi: 10.2215/CJN.06540810. Epub 2011 Jan 13. PMID 21233458
- [Background] Gheorghiade M, Niazi I, Ouyang J, Czerwiec F, Kambayashi J, Zampino M, Orlandi C; Tolvaptan Investigators. Vasopressin V2-receptor blockade with tolvaptan in patients with chronic heart failure: results from a double-blind, randomized trial. Circulation. 2003 Jun 3;107(21):2690-6. doi: 10.1161/01.CIR.0000070422.41439.04. Epub 2003 May 12. PMID 12742979
- [Background] Hauptman PJ, Zimmer C, Udelson J, Shoaf SE, Mallikaarjun S, Bramer SL, Orlandi C. Comparison of two doses and dosing regimens of tolvaptan in congestive heart failure. J Cardiovasc Pharmacol. 2005 Nov;46(5):609-14. doi: 10.1097/01.fjc.0000180899.24865.b6. PMID 16220067